CLINICAL TRIAL: NCT02815852
Title: RETROSPECTIVE ANALYSIS OF BREAST BIOPSIES IN WOMEN YOUNGER THAN 40 YEARS OLD
Acronym: RAD2016
Status: Completed | Type: Observational
Sponsor: Azienda U.S.L. 1 di Massa e Carrara (Other)
Responsible Party: Sponsor
Other Study IDs: Az.USLToscana Nord Ovest
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer in Women Under 40 Years Old
Keywords: breast cancer in women under 40 years old; biopsy; ultrasonography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Women under 40 years old with histological diagnosis of breast cancer — Evaluation of imaging characteristics (ultrasound, mammography and mammary MRI if available) of breast cancer with the corresponding histological reports and assess whether in women <40 years the typical imaging presentation pattern of malignancies observed in women> 40 years are confirmed.

SUMMARY:
The purpose of this study is to review retrospectively cases of breast cancer of the centers belonging to the BREST UNIT Tuscany North-West Wide Area and compare the imaging characteristics (ultrasound, mammography and mammary MRI if available) of breast cancer with the corresponding histological reports and assess whether in women <40 years the typical imaging presentation pattern of malignancies observed in women> 40 years are confirmed.

DETAILED DESCRIPTION:
Breast cancer is the most frequent cancer in women and the leading cause of death in women under 50 years in the USA. In Italy, the Pool Airtum 2007-2010 figures confirm that breast cancer, excluding skin cancers, is 29% of cancers diagnosed in women and the leading cause of death in women, for the regions in which are active the cancer registries . Among women, breast cancer ranks first in all age groups: represents 29% of deaths in women aged <49 years, 23% in women between 50 and 69 years and 16% between women aged> 70 years. The disease is uncommon before age 30 but the European Cancer registries have detected since 1990 an increased incidence of breast cancer in women before age 40. For this reason it can be important to start to verify the incidence of breast cancer before age 40 in the BREAST UNIT of the Tuscany North-West Wide Area (Versilia, Lucca and Massa-Carrara). Mammography, which is the reference examination for prevention in women after age 40, has not shown before this age evidence of efficacy. Ultrasound examination, complementary to mammography, is generally well tolerated but did not demonstrate efficacy in prospective studies as a screening in reducing mortality. MRI with intravenous contrast medium is considered the exam with higher sensitivity in identifying neoplastic lesions especially in young women. This study therefore aims to review retrospectively cases of breast cancer of the centers belonging to the BREST UNIT Tuscany North-West Wide Area to locate a number of cases to allow for a comparison on the imaging characteristics (ultrasound, mammography and mammary MRI if available) of breast cancer and assess whether in women <40 years the typical imaging presentation pattern of malignancies observed in women> 40 years are confirmed. In this study will be involved pathological anatomy of the BREAST UNIT Tuscany North-West Wide Area (Massa-Carrara, Versilia, Lucca); Radiology (Massa-Carrara, Versilia, Lucca); Clinical breast surgery / oncology / radiology of the three USL (Massa-Carrara, Versilia, Lucca) of the Tuscany North-West Wide Area. Data of patients diagnosed with breast cancer from 01/01/2009 to 31/12/2015 will be collected starting in july 2016 and the publication of results will take place by December 2016.Risk factors, genetic mutations, receptors status, tumor stage, therapies for NHL / LH and previous breast tumors will be analyzed as well. The data will be stratified by: age (<30 years, 30-35 years and 35-39 years), biological parameters on histology, stage at diagnosis and imaging features. Patients undergoing breast biopsy sampling represent an already select group who may be susceptible to information bias inherent risk factors: to reduce this bias will recover all the information about the risk factors for breast cancer. 2) operator-dependent variability of ultrasound images: will be taken into account in the data analysis, as well as different machines used in the various hospitals and diversity of the reporting method. 3) The patients for which it will not be possible to correct analysis of the data will be excluded, but the selection bias of patients will still be taken into account in the analysis of the data.The statistical analysis will be done in 1 month, and the results will be published by December 2016.

ELIGIBILITY:
Inclusion Criteria:

* Women aged <40 years with breast cancer diagnosis from 01/01/2009 to 31/12/2015 by imaging guided biopsy and / or histology of the surgical specimen extracted from the database of pathological anatomy afferent BREAST UNIT of Tuscany North-West Wide Area.

Exclusion Criteria:

* Women aged > 40 years with breast cancer diagnosis from 01/01/2009 to 31/12/2015 by imaging guided biopsy and / or histology of the surgical specimen extracted from the database of pathological anatomy afferent BREAST UNIT of Tuscany North-West Wide Area.
* Women aged <40 years with breast cancer diagnosis before 01/01/2009 of after 31/12/2015 by imaging guided biopsy and / or histology of the surgical specimen extracted from the database of pathological anatomy afferent BREAST UNIT of Tuscany North-West Wide Area.
* Patients with ultrasound examination and risk factors not available

Max Age: 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women aged <40 years with breast cancer diagnosis from 01/01/2009 to 31/12/2015 by imaging guided biopsy and / or histology of the surgical specimen extracted from the database of pathological anatomy afferent BREAST UNIT of Tuscany North-West Wide Area.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Compare the imaging features of benign and malignant mammary lesions in women <40 years with histological examinations to assess the correlatability between imaging morphology and histological characteristic of breast lesions. | September 2016
  It will be made a comparison between the radiological and histological reports of all patients with breast cancer diagnosis.

SECONDARY OUTCOMES:
Evaluate the incidence of malignant breast disease on total access to the Breast Unit of the Tuscany North-West Wide Area in patients <40 years | September 2016